CLINICAL TRIAL: NCT00504153
Title: A Phase II Study of Dasatinib (NSC 732517) in Previously-Treated Patients With Metastatic Colorectal Cancer
Brief Title: Dasatinib in Treating Patients With Previously Treated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00223; NCI-2009-00223 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCCRC-NCI-7786; CDR0000557036; 15431A (Other: University of Chicago); 7786 (Other: CTEP); N01CM62201 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Results first posted 2013-09-10 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2011-10

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Dasatinib

ARMS (1):
- Treatment (tyrosine Kinase Inhibitor) (Experimental): Patients receive oral dasatinib twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dasatinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: dasatinib
  Other Names: BMS-354825; Sprycel
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying dasatinib to see how well it works in treating patients with previously treated metastatic colorectal cancer. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the progression-free survival of patients with metastatic colorectal cancer who have progressed on or following two prior chemotherapy regimens and are then treated with dasatinib.

SECONDARY OBJECTIVES:

I. Determine the objective response rates in patients treated with dasatinib. II. Determine the overall survival of patients treated with dasatinib. III. Determine the toxicity in patients treated with dasatinib.

TERTIARY OBJECTIVES:

I. Determine the incidence of somatic mutations in c-src, c-yes, fyn, lck, hck, lyn, yrk and csk in archival primary and metastatic colorectal cancer tissues from these patients and to correlate this with clinical outcome.

II. Determine the incidence of total c-src and phosphorylated c-src expression in archival primary and metastatic colorectal cancer specimens from these patients, and to correlate this with clinical outcome.

III. Evaluate the effect of dasatinib on serum VEGF levels.

OUTLINE: This is a multicenter study. Patients receive oral dasatinib twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Blood is collected on days 1 (prior to the first dose of dasatinib) and 15 of course 1 for measurement of VEGF pre-and post-dasatinib administration. Archived tumor tissue (tumor or core biopsy; primary or metastatic lesion) is collected for identification of the incidence of somatic mutations and polymorphisms by polymerase chain reaction and electrophoresis and for measurement of total c-src and phosphorylated src expression by immunohistochemistry.

After completion of study treatment, patients are followed for at least 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed colorectal cancer

  * Metastatic disease
  * Not curable by surgical resection
  * Archival tumor tissue available
* Measurable disease, defined as at least one unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan

  * Measurable disease must be outside of a prior radiation port
* Documented disease progression either during or after prior chemotherapy treatment
* No more than 2 prior chemotherapy regimens in the adjuvant or metastatic setting

  * Prior chemotherapy regimens must have contained a fluoropyrimidine (e.g., fluorouracil or capecitabine), oxaliplatin, and irinotecan

    * Patients who received no prior adjuvant therapy must have received 2 prior chemotherapy regimens for metastatic disease (e.g., FOLFOX followed by FOLFIRI)
    * Patients who received prior adjuvant therapy with a fluoropyrimidine plus oxaliplatin must have received no more than 1 chemotherapy regimen for metastatic disease that must have contained irinotecan
    * VEGF or EGFR inhibitors with prior chemotherapy allowed
* No known brain metastases
* Life expectancy > 3 months
* ECOG performance status (PS) 0-2 or Karnofsky PS ≥ 60%
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST/ALT ≤ 2.5 times ULN (5 times ULN with liver metastases)
* Creatinine normal or creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to dasatinib
* No QTc prolongation, defined as a QTc interval ≥ 480 msecs (Bazett correction)
* No condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, or active peptic ulcer disease) that would impair ability to swallow and retain dasatinib tablets

  * Prior partial colectomy is not considered an exclusion factor
* No clinically significant cardiovascular disease including any of the following:

  * Myocardial infarction or ventricular tachyarrhythmia within the past 6 months
  * New York Heart Association class II -IV congestive heart failure
  * Major conduction abnormality (unless a cardiac pacemaker is present)
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * History of significant bleeding disorder (including congenital [e.g., von Willebrand's disease] or acquired [e.g., anti-factor VIII antibodies] disorders)
  * Large pleural effusions
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No currently active second malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix

  * Patients are not considered to have a currently active malignancy if they have completed therapy and have no evidence of recurrence for at least 5 years
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* At least 4 weeks since prior radiation therapy and recovered
* No prior surgical procedures affecting absorption
* No prior treatment with inhibitors of src, PDGFR, KIT, or EPHA2
* More than 1 week since prior and no concurrent medications or substances that are potent inhibitors or inducers of CYP3A4
* More than 1 week since prior and no concurrent medications that inhibit platelet function (e.g., aspirin, dipyridamole, epoprostenol, eptifibatide, clopidogrel, cilostazol, abciximab, ticlopidine, or any non-steroidal anti-inflammatory drug)
* More than 1 week since prior and no concurrent agents that are generally accepted to have a risk of causing Torsades de Pointes, including quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide, erythromycins, clarithromycin, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, or lidoflazine
* No concurrent anticoagulants (e.g., warfarin, heparin/low molecular weight heparin [e.g., danaparoid, dalteparin, tinzaparin, or enoxaparin])
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent grapefruit or grapefruit juice
* No other concurrent investigational agents or commercial agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasatinib (Tyrosine Kinase Inhibitor): Patients receive oral dasatinib twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dasatinib (Tyrosine Kinase Inhibitor)
Started | 19
Completed | 13
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 4
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib (Tyrosine Kinase Inhibitor)
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 64 [34 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate
Description: Progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Patients who are still alive and have not progressed will be censored at the date of the last negative examination. A Simon (1989), optimal, two-stage design will be employed. The progression-free survival count will be the proportion of subjects who are alive and progression-free at 4 months.
Time Frame: From the start of treatment to the time of disease progression or death from any cause, assessed at 4 months after completion of treatment (i.e., up to 12 months.)
Measure: Number; unit: percentage of participants
Arm/Group | Dasatinib (Tyrosine Kinase Inhibitor)
Number analyzed (Participants) | 19
percentage of participants | 5.3

2. Secondary Outcome: Response Rate (RR) (Complete or Partial Responders)
Description: Response will be evaluated in this study using the new international criteria proposed by the RECIST Committee. The response rate is the proportion of subjects who experienced a complete or partial response.
Time Frame: Every 2 courses, assessed up to 8 weeks after completion of study treatment (i.e., up to 10 months)
Measure: Number; unit: percentage of participants
Arm/Group | Dasatinib (Tyrosine Kinase Inhibitor)
Number analyzed (Participants) | 19
percentage of participants | 0

3. Secondary Outcome: Incidence of Somatic Mutations
Description: Multivariable analysis of progression-free survival duration will be performed using the Cox (1972) regression model to evaluate the prognostic value of somatic mutations. For the mutational analysis endpoints, genetic mutations will also be correlated with drug activity via Fisher's exact test for comparisons of responders with non-responders and for comparison of patients progression-free and 4 months vs. those with early progression or death
Time Frame: 1 year
Population: This outcome was not assessed for any of the patients.
Arm/Group | Dasatinib (Tyrosine Kinase Inhibitor)
Number analyzed (Participants) | 0

4. Secondary Outcome: Association Between the Incidence of Total C-src and Phosphorylated C-src Expression and Response
Description: Examined by comparing expression in those who have an objective response versus those who do not and in those with and without disease progression at 4 months using Fisher's exact test.
Time Frame: 4 months
Population: This outcome was not assessed for any of the patients.
Arm/Group | Dasatinib (Tyrosine Kinase Inhibitor)
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Plasma Vascular Endothelial Growth Factor (VEGF) Levels Over 15 Days
Description: Changes of VEGF will be correlated with response rates and 4-month progression-free survival utilizing the Wilcoxon rank-sum test.
Time Frame: At baseline and day 15
Population: This outcome was not assessed for any of the patients.
Arm/Group | Dasatinib (Tyrosine Kinase Inhibitor)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Patients were followed for approximately 2 months after study treatment, approximately 6 months.
Description: All serious adverse events are reported here. The non-serious adverse (NSAE) events report includes those NSAEs assessed at grade 3 or higher.
Arm/Group | Dasatinib (Tyrosine Kinase Inhibitor)
Serious Adverse Events (participants affected / at risk) | 10/19
Other Adverse Events (participants affected / at risk) | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (Tyrosine Kinase Inhibitor) (N=19)
Abdominal pain (General disorders) | 2 — Pain in the abdominal region
Acute kidney injury (Renal and urinary disorders) | 1 — Acute kidney injury (AKI), previously called acute renal failure (ARF), is a rapid loss of kidney function.
Anorexia (Gastrointestinal disorders) | 1 — Anorexia is the decreased sensation of appetite.
Ascites (Gastrointestinal disorders) | 1 — Ascites is a gastroenterological term for an accumulation of fluid in the peritoneal cavity.
Blood infection (Blood and lymphatic system disorders) | 1 — Blood infection with normal ANC or Grade 1 or 2 neutrophils
Creatinine increased (Metabolism and nutrition disorders) | 1 — Increased levels of creatinine
Dehydration (Gastrointestinal disorders) | 2 — Dehydration (hypohydration) is the excessive loss of body water, with an accompanying disruption of metabolic processes.
Diarrhea (Gastrointestinal disorders) | 1 — Diarrhea is the condition of having three or more loose or liquid bowel movements per day.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 — Shortness of breath
Fever (General disorders) | 1 — Fever is characterized by an elevation of body temperature above the normal range of 36.5-37.5 °C (97.7-99.5 °F) due to an increase in the temperature regulatory set-point
Gastritis (Gastrointestinal disorders) | 1 — Gastritis is an inflammation of the lining of the stomach.
Headache (General disorders) | 1 — A headache or cephalalgia is pain anywhere in the region of the head or neck.
Hyperkalemia (Metabolism and nutrition disorders) | 1 — Hyperkalemia refers to the condition in which the concentration of the electrolyte potassium (K+) in the blood is elevated.
Hypokalemia (Metabolism and nutrition disorders) | 1 — Hypokalemia refers to the condition in which the concentration of potassium (K+) in the blood is low.
Hyponatremia (Metabolism and nutrition disorders) | 1 — Hyponatremia is an electrolyte disturbance in which the sodium ion concentration in the serum is lower than normal.
Hypotension (Cardiac disorders) | 2 — Hypotension is low blood pressure, especially in the arteries of the systemic circulation
Nausea (Gastrointestinal disorders) | 2 — Nausea is a sensation of unease and discomfort in the upper stomach with an involuntary urge to vomit.
Pancreatitis (Hepatobiliary disorders) | 1 — Pancreatitis is an inflammation of the pancreas
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 — Pleural effusion is excess fluid that accumulates between the two pleural layers, the fluid-filled space that surrounds the lungs.
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 — Pneumonitis or pulmonitis is a general term that refers to inflammation of lung tissue.
Syncope (General disorders) | 1 — Syncope (fainting) is a transient loss of consciousness and postural tone, characterized by rapid onset, short duration, and spontaneous recovery.
Urinary tract infection (Infections and infestations) | 2 — A urinary tract infection (UTI) (also known as acute cystitis or bladder infection) is an infection that affects part of the urinary tract.
Ventricular fibrillation (Cardiac disorders) | 1 — Ventricular fibrillation (V-fib or VF) is a condition in which there is uncoordinated contraction of the cardiac muscle of the ventricles in the heart, making them quiver rather than contract properly.
Vomiting (Gastrointestinal disorders) | 2 — Vomiting (known medically as emesis and informally as throwing up and numerous other terms) is the forceful expulsion of the contents of one's stomach through the mouth and sometimes the nose.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (Tyrosine Kinase Inhibitor) (N=19)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 — Increased levels of alanine aminotransferase, indicative of liver damage or disease.
Alkaline phosphatase (ALP) increased (Metabolism and nutrition disorders) | 1 — Increased levels of Alkaline phosphatase
Anemia (Blood and lymphatic system disorders) | 2 — Anemia is a decrease in number of red blood cells (RBCs) or less than the normal quantity of hemoglobin in the blood.
Anorexia (Gastrointestinal disorders) | 1 — Anorexia is the decreased sensation of appetite.
Aspartate aminotransferase (AST) increased (Metabolism and nutrition disorders) | 1 — Increased levels of aspartate aminotransferase (AST)
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 — Increased levels of bilirubin in the blood
Blood infection (Infections and infestations) | 1 — Blood infection with normal absolute neutrophil count (ANC) or Grade 1 or 2 neutrophils
Duodenal stenosis (Gastrointestinal disorders) | 1 — A rare birth defect where a portion of the small intestine is narrowed which prevents the stomach contents from flowing through at a normal rate.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 — Shortness of breath
Fatigue (General disorders) | 3 — Fatigue (also called exhaustion, tiredness, lethargy, languidness, languor, lassitude, and listlessness) is a subjective feeling of tiredness which is distinct from weakness, and has a gradual onset.
Hemorrhoids (Gastrointestinal disorders) | 1 — Hemorrhoids, also called piles, are swollen and inflamed veins in your anus and lower rectum.
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 — Hypoalbuminemia is a medical condition where levels of albumin in blood serum are abnormally low.
Hypoglycemia (Metabolism and nutrition disorders) | 1 — Hypoglycemia is an abnormally diminished content of glucose in the blood.
Hypokalemia (Metabolism and nutrition disorders) | 1 — Hypokalemia refers to the condition in which the concentration of potassium (K+) in the blood is low.
Hyponatremia (Metabolism and nutrition disorders) | 1 — Hyponatremia is an electrolyte disturbance in which the sodium ion concentration in the serum is lower than normal.
INR increased (Blood and lymphatic system disorders) | 1 — Above normal international normalized ratio (INR)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 — Lymphocyte count decreased
Peripheral sensory neuropathy (Nervous system disorders) | 1 — Inflammation or degeneration of the sensory nerves.
Rectal pain (Gastrointestinal disorders) | 1 — Rectal pain is the symptom of pain in the area of the rectum.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less